CLINICAL TRIAL: NCT03275298
Title: Epidemiological Strategy and Medical Economic (ESME) Research Program / Academic Real World Database : Evolution of the Therapeutic Care in Ovarian Cancer Across the French Comprehensive Cancer Centers From 2011
Brief Title: Evolution of the Therapeutic Care in Ovarian Cancer From 2011
Acronym: ESME OC
Status: Suspended | Type: Observational
Why Stopped: enrolment temporariliy stopped for budget considerations
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Other Study IDs: ESME OC
Record Dates: First submitted 2017-06-27; First posted 2017-09-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; observational study; survival; real world data; real life setting
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer cohort: Any female treated for ovarian cancer in a French comprehensive cancer centers

SUMMARY:
The ESME Ovarian Cancer database is a multi-center real life database using a retrospective data collection process in 18 French Comprehensive Cancer Center (FCCC) over 20 sites). This database compiles data from existing data available from patient's electronic medical records (EMR).

DETAILED DESCRIPTION:
This database compiles data from existing data available from patient's electronic medical records (EMR) and integrates data from non-structured ans structured sources.

The database includes data related to patient demographics, tumor characteristics (diagnosis, histology, relapses, metastatic disease, etc.), treatments (dates, INN, route of administration, treatment protocols, reason for termination, etc.), and clinical events. Data is collected at each participating site by technicians who are specifically trained for the project using an electronic data collection (eDC) tool.

Data imported into the final database are controlled, recoded, and harmonized before import according to the data management plan. All coding procedures are predefined by the data manager. There is no transmission of individual data; all data are centralized within each center using a shared anonymous format. All data is exclusively obtained retrospectively; no attempts are made to recover non available data from the patient's medical record by contacting healthcare providers or patients.

ESME OC database aims to be a clinical and therapeutic database centralizing existing and available data from different sources used in the participating hospitals. Data do not contain any personal data on patients. In compliance with the authorization delivered by the French Data Protection agency to Unicancer, only aggregated statistical reports and publication are released.

ELIGIBILITY:
Inclusion criteria :

* 18 years old female
* Female who received surgery, chemotherapy, targeted therapy, immunotherapy, radiation therapy, diagnostic procedure, other specific therapeutic procedure) for ovarian cancer in a French Comprehensive Cancer Center.

Exclusion criteria : None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive females treated for an ovarian cancer in a French Comprehensive Cancer Center over the selection period.
Sampling Method: Non-Probability Sample
Enrollment: 13331 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Describe the evolution of therapeutic care in ovarian cancer across the French comprehensive cancer centers | baseline
  Patient characteristics, tumor characteristics and treatment patterns

SECONDARY OUTCOMES:
Describe the impact of therapeutic strategies on survival criteria | From date of diagnosis or first treatment until the date of date of death from any cause. Follow up until 2022.
  Overall survival

OTHER OUTCOMES:
Describe the impact of therapeutic strategies on survival criteria | From date of diagnosis or first treatment until the date of first documented progression or date of death from any cause. Follow up until 2022.
  Progression free survival

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer Montpellier / Val d'Aurelle, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - Institut de cancérologie de l'Ouest - René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
In accordance with ethical and legal requirements related to the ESME Data Warehouse, individual data from the ESME databases cannot be made available outside Unicancer secured servers.

REFERENCES:
- [Result] Romeo, C, P Meeus, M Rodrigues, E Leblanc, A Floquet, P Pautier, F Marchal, et al. " EP967 Natural history of patients with BRCA-mutated high grade epithelial ovarian cancer (HGEOC) before the era of PARP inhibitors maintenance in 1st line treatment ". In ePoster, A513.3-A513. BMJ Publishing Group Ltd, 2019. https://doi.org/10.1136/ijgc-2019-ESGO.1013.
- [Result] De Nonneville A, Zemmour C, Frank S, Joly F, Ray-Coquard I, Costaz H, Classe JM, Floquet A, De la Motte Rouge T, Colombo PE, Sauterey B, Leblanc E, Pomel C, Marchal F, Barranger E, Savoye AM, Guillemet C, Petit T, Pautier P, Rouzier R, Gladieff L, Simon G, Courtinard C, Sabatier R. Clinicopathological characterization of a real-world multicenter cohort of endometrioid ovarian carcinoma: Analysis of the French national ESME-Unicancer database. Gynecol Oncol. 2021 Oct;163(1):64-71. doi: 10.1016/j.ygyno.2021.07.019. Epub 2021 Jul 19. PMID 34294414
- [Result] Rodrigues M, Joly F, Ray-Coquard I, Costaz H, Classe JM, Floquet A, De la Motte Rouge T, Colombo PE, Provensal Gross M, Leblac E, Pomel C, Marchal F, Barranger E, Savoye AM, Guillemet C, Petit T, Pautier P, Rouzier R, Courtinard C, Gladieff L. Real-world clinical outcomes of patients with de novo advanced high-grade epithelial ovarian cancer eligible to niraparib maintenance in France. ESMO Congress, September 16-21, 2021 [ePoster 746P] DOI:https://doi.org/10.1016/j.annonc.2021.08.1188
- [Result] Thomas QD, Boussere A, Classe JM, Pomel C, Costaz H, Rodrigues M, Ray-Coquard I, Gladieff L, Rouzier R, Rouge TM, Gouy S, Barranger E, Sabatier R, Floquet A, Marchal F, Guillemet C, Polivka V, Martin AL, Colombo PE, Fiteni F. Optimal timing of interval debulking surgery for advanced epithelial ovarian cancer: A retrospective study from the ESME national cohort. Gynecol Oncol. 2022 Oct;167(1):11-21. doi: 10.1016/j.ygyno.2022.08.005. Epub 2022 Aug 13. PMID 35970603
- [Result] Bini M, Quesada S, Meeus P, Rodrigues M, Leblanc E, Floquet A, Pautier P, Marchal F, Provansal M, Campion L, Causeret S, Gourgou S, Ray-Coquard I, Classe JM, Pomel C, De La Motte Rouge T, Barranger E, Savoye AM, Guillemet C, Gladieff L, Demarchi M, Rouzier R, Courtinard C, Romeo C, Joly F. Real-World Data on Newly Diagnosed BRCA-Mutated High-Grade Epithelial Ovarian Cancers: The French National Multicenter ESME Database. Cancers (Basel). 2022 Aug 21;14(16):4040. doi: 10.3390/cancers14164040. PMID 36011033
- [Result] Brouillard-Saby F, Saint-Martin C, Ray-Coquard I, Gladieff L, Pomel C, Colombo PE, Classe JM, Chevrier M, Joly F, De la Motte Rouge T, Floquet A, Sabatier R, Barranger E, Costaz H, Leblanc E, Marchal F, Pautier P, Bosquet L, Rodrigues M. Efficacy of chemotherapy according to BRCA status in patients with high-grade serous ovarian carcinoma at first platinum-sensitive relapse. Int J Gynecol Cancer. 2023 Apr 3;33(4):577-584. doi: 10.1136/ijgc-2022-003993. PMID 36631150
- [Derived] Rippstein N, Zemmour C, Rodrigues M, Ray-Coquard I, Gladieff L, Pautier P, Frenel JS, Costaz H, Lebreton C, Pomel C, Colombo PE, Marchal F, Guillemet C, de la Motte Rouge T, Eberst L, Bosquet L, Deluche E, Sabatier R. PARP inhibitors as maintenance therapy in ovarian cancer after platinum-sensitive recurrence: real-world experience from the Unicancer network. Oncologist. 2025 May 8;30(5):oyaf075. doi: 10.1093/oncolo/oyaf075. PMID 40349134